CLINICAL TRIAL: NCT03644953
Title: Hydroxyurea and Transfusion: Pilot Study of Combination Therapy for Patients With Sickle Cell Anemia
Brief Title: Hydroxyurea and Transfusion
Acronym: HAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Robert Nickel, Principal Investigator, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00010541
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Sickle Cell Disease
Keywords: Hydroxyurea; Transfusion
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, open label study of combination hydroxyurea and simple chronic transfusion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hydroxyurea and Transfusion (HAT) (Experimental): Combination hydroxyurea and simple chronic transfusion therapy
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — Participants will be started on hydroxyurea 20 ± 2.5 mg/kg/day in addition to continuing simple chronic transfusion every 4 weeks ± 1 week. Hydroxyurea will be dose escalated to achieve a HAT target dose (HAT-TD). Hydroxyurea will be increased by 5 mg/kg/day after 8 weeks of a dose if HAT-TD is not achieved (maximum daily dose 2,000 mg). After HAT-TD has been achieved, minor dose increases may occur if subject grows a significant amount to maintain the same mg/kg dose.

SUMMARY:
This study will prospectively investigate the feasibility, safety, and transfusion requirements of adding hydroxyurea to simple chronic transfusions for patients with sickle cell anemia already on chronic transfusions.

DETAILED DESCRIPTION:
This is a single-arm, prospective study of hydroxyurea added to simple chronic transfusions, combination treatment termed hydroxyurea and transfusion (HAT). The primary objective of the study is to determine the feasibility of HAT for patients with sickle cell anemia (SCA) currently being treated only with simple transfusions for stroke prevention. Secondary objectives include: to evaluate the safety of HAT and to determine if HAT decreases transfusion requirements in this patient population. Exploratory objectives include: to evaluate with HAT changes in pre-transfusion laboratories and biomarkers of cerebrovascular disease progression, and to describe changes on brain imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SCA (Hb SS or Sβ0 thalassemia).
2. On simple chronic transfusion therapy for stroke prevention (primary or secondary prevention) for ≥1 year with no plans to stop simple chronic transfusion in the next year.

Exclusion Criteria:

1. Poor adherence to simple transfusion regimen as defined by having an HbS >45% at any time in the last year AND a transfusion interval >5 weeks.
2. Treatment with hydroxyurea in the 12 months prior to study enrollment.
3. Abnormal initial laboratory values (temporary exclusions):

   1. Absolute neutrophil count <1.5 x 10^9/L
   2. Platelet count <100 x 10^9/L
   3. Serum creatinine more than twice upper limit for age
4. Pregnancy or unwillingness to use a medically acceptable form of contraception if sexually active.

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Recruitment ratio | 1 year
  number of participants who enroll on the study / total number of eligible subjects
Retention ratio | 1 year
  number participants who remain on study 1 year after HAT target dose / total number enrolled participants
Hydroxyurea adherence ratio | 1 year
  (hydroxyurea amount dispensed - amount returned) / prescribed amount between visits

SECONDARY OUTCOMES:
Proportion of subjects who develop an hemoglobin (Hb) S >45% AND an Hb >11.0 g/dL | 1 year
  incidence of above safety event will be monitored closely throughout the trial
Volume of red blood cells transfused per patient weight | 1 year
  measure to evaluate the transfusion requirement of HAT

CONTACTS AND LOCATIONS:
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No